CLINICAL TRIAL: NCT00822770
Title: G-CSF and Plerixafor With Busulfan and Fludarabine for Allogeneic Stem Cell Transplantation for Myeloid Leukemias
Brief Title: Plerixafor and Granulocyte Colony-stimulating Factor (G-CSF) With Busulfan, Fludarabine and Thymoglobulin
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0772
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Results first posted 2014-07-16 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-09

CONDITIONS: Stem Cell Transplantation; Leukemia
Keywords: Blood Stem Cell Transplantation; Bone Marrow Transplantation; Bone Marrow Cell Transplantation; Stem Cell Transplantation; Allogeneic Hematopoietic Transplantation; Advanced Myeloid Leukemia; Acute Myeloid Leukemia; AML; Myelodysplastic syndrome; MDS; Chronic Myeloid Leukemia; CML; Graft Versus Host Disease; GVHD; ATG; Busulfan; Busulfex™; Myleran®; Filgrastim; Neupogen; Fludarabine; Fludarabine Phosphate; Fludara™; G-CSF; Plerixafor; Antithymocyte globulin; Thymoglobulin
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Graft vs Host Disease | interventions — plerixafor; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine; fludarabine phosphate; Busulfan; Bone Marrow Transplantation; thymoglobulin; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase I (Experimental): ATG + Plerixafor (AMD3100) + G-CSF (Filgrastim) + Fludarabine + Busulfan + Allogeneic blood stem cell transplant
  Interventions: Drug: Plerixafor; Drug: Filgrastim; Drug: Fludarabine; Drug: Busulfan; Procedure: Allogeneic blood stem cell transplant; Drug: ATG (Thymoglobulin)
- Phase II (Experimental): ATG + MTD Plerixafor (AMD3100) + G-CSF (Filgrastim) + Fludarabine + Busulfan + Allogeneic blood stem cell transplant
  Interventions: Drug: Plerixafor; Drug: Filgrastim; Drug: Fludarabine; Drug: Busulfan; Procedure: Allogeneic blood stem cell transplant; Drug: ATG (Thymoglobulin)

INTERVENTIONS:
Drug: Plerixafor — Phase I: Starting dose of 0 (escalating doses 80, 160, 240 mcg/kg) given daily subcutaneously in abdomen for 4 doses.
  Phase II: Maximum Tolerated Dose (MTD) as determined in Phase I
  Other Names: AMD3100
Drug: Filgrastim — Dose of 10 mcg/kg subcutaneous injection beginning on day -9 daily for 6 days.
  Other Names: G-CSF; Neupogen
Drug: Fludarabine — Dose of 40 mg/m^2 beginning on Day -6 for four consecutive days.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Busulfan — Dose of 130 mg/m^2 for four consecutive days, immediately after completion of Fludarabine.
  Other Names: Busulfex™; Myleran®
Procedure: Allogeneic blood stem cell transplant — Stem Cell Infusion (Bone marrow or PBPC)
  Other Names: Bone Marrow Transplantation; Blood Stem Cell Transplantation
Drug: ATG (Thymoglobulin) — Dose(s) of 0.5 mg/kg on day -3; of 1.5 mg/kg on day -2; and of 2 mg/kg on day -1. Given only to patients with unrelated donors.
  Other Names: Antithymocyte globulin

SUMMARY:
The goal of this clinical research study is to learn about the safety of AMD3100 (plerixafor) and G-CSF (filgrastim) in combination with fludarabine, busulfan, and an allogeneic blood stem cell transplant. This treatment will be studied in patients with acute myeloblastic leukemia (AML), myelodysplastic syndromes (MDS), or Chronic myelogenous leukemia (CML).

DETAILED DESCRIPTION:
The Study Treatment:

Fludarabine is a chemotherapy drug that is designed to make cancer cells less able to repair damaged DNA (the genetic material of cells). This may increase the likelihood of the cells dying.

Busulfan is a chemotherapy drug that is designed to bind to DNA, which may cause cancer cells to die. It is commonly used in stem cell transplants.

Plerixafor and filgrastim are designed to cause cancer cells to move from the bone marrow into the blood stream. This may help to make the cancer cells more sensitive to being killed by the chemotherapy.

An "allogeneic" (from a donor) stem cell transplant is designed to help the recipient's body attack the cancer cells that may remain in the body after chemotherapy.

Study Groups and Plerixafor Dose Levels:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 4 groups of 3 participants will be enrolled in the Phase I portion of the study, and up to 48 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of plerixafor you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of plerixafor. Each new group will receive a higher dose of plerixafor than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of plerixafor is found.

If you are enrolled in Phase II, you will receive plerixafor at the highest dose that was tolerated in the Phase I portion.

In this study, plerixafor is the only study drug where different dose levels are being tested and compared.

Drug Administration Before the Transplant:

You will receive your first dose of filgrastim on Day -9. (Day -9 means 9 days before the stem cell transplant, which will occur on Day 0).

Filgrastim is injected under the skin once a day from Day -9 through Day -4. Plerixafor is injected under the skin once a day from Day -7 through Day -4. The plerixafor injections will occur 8 hours before the fludarabine and busulfan chemotherapy.

The fludarabine and busulfan will be given by vein through a central venous catheter (CVC). A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

Fludarabine is given once a day from Day -6 through Day -3, over 1 hour each time. On these same days, busulfan will be given after the fludarabine, over 3 hours.

You will also receive tacrolimus in order to lower the risk of graft vs. host disease (GVHD). GVHD is a disease that occurs when the donor's immune cells react against the recipient's body, attacking the recipient's cells and tissues.

Starting on Day -2, tacrolimus will be given as a continuous (non-stop) infusion through the CVC. When the study doctor decides it seems safe, you will begin taking tacrolimus by mouth instead, for as long as the study doctor decides is necessary.

If your stem cell donor is not someone who is related to you, you will receive antithymocyte globulin (ATG) through the CVC once a day from Day -3 through Day -1. On Day -3, it will be given over at least 6 hours. On Days -2 and -1, it will be given over at least 4 hours. This drug is given in order to weaken your immune system in order to lower the risk of your immune system rejecting the transplanted cells.

Blood Tests Before the Transplant:

If you are in the Phase I part of this study, the following blood samples will be drawn and are not optional. Eight total blood samples (about 1 1/2 teaspoons each) will be drawn daily with your routine morning labs beginning before your first dose of study therapy (or Day -9) through Day -3. These samples will be used for research purposes, to study how the chemotherapy drugs and transplant may affect your normal cells and cancerous cells.

If you are in the Phase II part of the study the following blood samples are optional and if you agree, eight total blood samples (about 1 1/2 teaspoons each) will be drawn daily beginning before your first dose of study therapy (or Day -9) through Day -3. These samples will be used for research purposes, to study how the chemotherapy drugs and transplant may affect your normal cells and cancerous cells.

Stem Cell Transplant:

On Day 0, after 2 days of rest from chemotherapy, the donor's stem cells will be given to you by vein (through the CVC). This should take about 30-60 minutes.

Drug Administration After the Transplant:

In addition to continuing to receive tacrolimus to lower the risk of GVHD (as described above), after the transplant you will also receive methotrexate to lower the risk of GVHD. Methotrexate will be given by vein, through the CVC, over 15 minutes on Days 1, 3, and 6. It will also be given on Day 11 if your stem cell donor is someone who is not related to you.

Once a day, starting at 1 week after the transplant, you will receive filgrastim as an injection under your skin. These daily injections will continue until your blood counts recover.

Reasons for Stopping the Study Treatment Early:

If you experience intolerable side effects or the disease gets worse during study treatment, you will be taken off the study treatment.

Other Procedures After the Transplant:

You will remain in the hospital until your blood counts recover (usually about 4 weeks after the transplant). You will continue being monitored for any infections and transplant-related side effects for at least 100 days after the transplant.

At 1, 3, 6, and 12 months after the transplant, you will have blood tests (about 3 tablespoons) and bone marrow biopsies performed to check the status of the disease.

Length of Study Participation:

Your active participation in this study will be over at 12 months after the transplant. The study staff will continue to contact your local doctor regularly from then on. The purpose is to check the status of the disease and see how you are doing.

Up to 72 patients will take part in this study. All will be enrolled at The University of Texas (UT) MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age >/=18 to </= 65 years.
2. Diagnosis of AML in first or greater remission, first or subsequent relapse, or primary induction failure; MDS with intermediate or high risk International Prognostic Scoring System (IPSS) score having failed to respond or recurred after chemotherapy; in remission or having active disease after treatment; AML arising from MDS; or CML which has failed to respond to imatinib or other tyrosine kinase inhibitor and has had >5% blasts in the blood or bone marrow. Patients receiving second transplants after relapse are considered in the relapse group.
3. White Blood Count (CBC) </= 20 * 10^9/l.
4. Patients should have a histocompatible, related or unrelated volunteer donor available. A histocompatible donor is defined as HLA matched related donor or an unrelated donor matched for HLA- A, B, C, and DR antigens by high-resolution DNA techniques.
5. Zubrod performance status 0 or 1, or Karnofsky performance status 90-100%.
6. Left ventricular ejection fraction >/= 45 %. No uncontrolled arrhythmias or uncontrolled symptomatic cardiac disease.
7. No symptomatic pulmonary disease. Forced expiratory volume in 1 s (FEV1), forced vital capacity (FVC) and diffusion capacity of carbon monoxide (DLCO) >/= 50 % of expected, corrected for hemoglobin.
8. Serum creatinine </=1.5 mg/dl.
9. Serum glutamic pyruvic transaminase (SGPT) </= 200 IU/ml unless related to the malignancy.
10. Total serum bilirubin </=1.5 mg/dl (unless Gilbert's syndrome) and alkaline phosphatase </=2.5 times laboratory standard upper limit of normal (ULN).
11. Patient or patient's legal representative able to sign informed consent.

Exclusion Criteria:

1. History of HIV positive.
2. Positive Beta human chorionic gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization.
3. Pleural/pericardial effusion or ascites estimated >/= 1 liter.
4. Uncontrolled infection, not responding to appropriate antimicrobial agents after seven days of therapy.
5. History of acute hepatitis, chronic active hepatitis or cirrhosis.
6. Patients with class 3 or 4 angina (New York Heart Association (NYHA) criteria).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2009-01; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Konopleva, MD, PhD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 2, 2009 to February 1, 2012. All recruitment done at the University of Texas MD Anderson Cancer Center.
Groups:
- Phase I Plerixafor + G-CSF: Plerixafor (AMD3100) Starting dose of 0 (escalating doses 80, 160, 240 mcg/kg) given daily subcutaneously in abdomen for 4 doses + Thymoglobulin (ATG) 0.5 mg/kg on day -3; 1.5 mg/kg on day -2; & 2 mg/kg on day -1. Given only to patients with unrelated donors + G-CSF (Filgrastim) 10 mcg/kg subcutaneous injection beginning on day -9 daily for 6 days + Fludarabine 40 mg/m^2 beginning on Day -6 for four consecutive days + Busulfan 130 mg/m^2 for four consecutive days, immediately after completion of Fludarabine + Allogeneic blood stem cell transplant of Stem Cell Infusion (Bone marrow or PBPC)
- Phase II Plerixafor 240 mcg/kg + G-CSF: Plerixafor Phase I Maximum Tolerated Dose (MTD) 240 mcg/kg daily for 4 days starting Day -7 + ATG 0.5 mg/kg day -3; 1.5 mg/kg on day -2; & 2 mg/kg on day -1 only for participants with unrelated donors + G-CSF 10 mcg/kg subcutaneous injection beginning day -9 daily for 6 days + Fludarabine 40 mg/m^2 beginning on Day -6 for four consecutive days + Busulfan 130 mg/m^2 for 4 consecutive days, immediately after completion of Fludarabine + Allogeneic blood stem cell transplant.
Period: Overall Study
Arm/Group | Phase I Plerixafor + G-CSF | Phase II Plerixafor 240 mcg/kg + G-CSF
Started | 18 | 29
Completed | 15 | 28
Not Completed | 3 | 1
Not completed — Not treated | 1 | 0
Not completed — Complication/Incomplete treatment | 1 | 0
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Plerixafor + G-CSF | Phase II Plerixafor 240 mcg/kg + G-CSF | Total
Number analyzed (Participants) | 18 | 29 | 47
Age, Continuous [Median (Full Range); unit: years] | 58 [41 to 65] | 53 [25 to 65] | 55 [25 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 17 | 26
  Male | 9 | 12 | 21
Region of Enrollment [Number; unit: participants]
  United States | 18 | 29 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 4 Dose Limiting Toxicity to Determine Maximum Tolerated Dose (MTD) Plerixafor
Description: Phase I determination of MTD dose of Plerixafor in combination with a fixed dose of Filgrastim where dose limiting toxicity defined as any grade 4 non-hematologic toxicity observed within 28 days from Day 0 (day of transplant).
Time Frame: 28 day cycle (Plerixafor Day -7 to Day -4)
Population: Two participants of 18 registered left the study without receiving Plerixafor treatment and there were not available for MTD analysis.
Measure: Number; unit: participants
Groups:
- Phase I Plerixafor + G-CSF: ATG + Plerixafor (AMD3100) + G-CSF (Filgrastim) + Fludarabine + Busulfan + Allogeneic blood stem cell transplant
  Allogeneic blood stem cell transplant : Stem Cell Infusion (Bone marrow or PBPC)
  Filgrastim : Dose of 10 mcg/kg subcutaneous injection beginning on day -9 daily for 6 days.
  Fludarabine : Dose of 40 mg/m^2 beginning on Day -6 for four consecutive days.
  ATG (Thymoglobulin) : Dose(s) of 0.5 mg/kg on day -3; of 1.5 mg/kg on day -2; and of 2 mg/kg on day -1. Given only to patients with unrelated donors.
  Busulfan : Dose of 130 mg/m^2 for four consecutive days, immediately after completion of Fludarabine.
  Plerixafor : Phase I: Starting dose of 0 (escalating doses 80, 160, 240 mcg/kg) given daily subcutaneously in abdomen for 4 doses.
Arm/Group | Phase I Plerixafor + G-CSF
Number analyzed (Participants) | 16
participants
  0 mcg/kg daily | 1
  80 mcg/kg daily | 4
  160 mcg/kg daily | 7
  240 mcg/kg daily | 4

2. Secondary Outcome: Number of Participants Alive With no Disease Progression at Time of Allo Transplant
Description: In Phase II portion of study, number of participants with treatment failure defined as either disease recurrence or death, measured from start of treatment to allo transplant at Day 0.
Time Frame: Baseline till transplant, Day -9 to Day 0, to 10 days
Population: Participants treated in the Phase 1 portion of the trial at the selected MTD dose were counted toward the maximum subgroup sample in Phase 2, therefore four of Phase I participants were included having received the MTD Plerixafor dose; however, one late participant in Phase 2 was not evaluable for the outcome.
Measure: Number; unit: percentage of participants
Groups:
- Overall Study: Plerixafor + G-CSF: Plerixafor escalating doses 0, 80, 160, 240 mcg/kg or MTD 240 mcg/kg given daily subcutaneously in abdomen for 4 doses + Thymoglobulin (ATG) 0.5 mg/kg on day -3; 1.5 mg/kg on day -2; & 2 mg/kg on day -1. Given only to patients with unrelated donors + G-CSF (Filgrastim) 10 mcg/kg subcutaneous injection beginning on day -9 daily for 6 days + Fludarabine 40 mg/m^2 beginning on Day -6 for four consecutive days + Busulfan 130 mg/m^2 for four consecutive days, immediately after completion of Fludarabine + Allogeneic blood stem cell transplant of Stem Cell Infusion (Bone marrow or PBPC)
Arm/Group | Overall Study: Plerixafor + G-CSF
Number analyzed (Participants) | 32
percentage of participants
  Participants in | 16
  Participants not in Complete Remission | 16

3. Secondary Outcome: Engraftment Response Rate: Number of Transplanted Participants With Complete Chimerism at Day 30
Description: Number of participants with complete chimerism at day 30 where defined as: Engraftment: first day of three (3) consecutive days that Absolute neutrophil count (ANC) exceeds 0.5 X 109/L. Subsequent chimerism studies must demonstrate the presence of donor derived cells. Graft Failure: failure to achieve an ANC >0.5 X 109/L for 3 consecutive days within 28 days after transplantation or a decline of ANC <0.5 x 109/L for three consecutive days after initial documented engraftment unless this is correlated with progression / recurrence of the underlying malignancy.
Time Frame: 30 Days post engraftment
Population: There were 39 participants receiving first transplants for acute myeloid leukemia (AML)/myelodysplastic syndrome (MDS) of both Phase I and Phase II who received MTD dose and allo transplant thus were evaluable for outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study: Plerixafor + G-CSF
Number analyzed (Participants) | 39
Participants | 32

ADVERSE EVENTS:
Time Frame: The active treatment period defined as study entry through Stem Cell Transfusion Day +28, follow up defined as Transfusion Day +29 through Day +100.
Groups:
- Phase I Plerixafor + G-CSF: ATG + Plerixafor (AMD3100) + G-CSF (Filgrastim) + Fludarabine + Busulfan + Allogeneic blood stem cell transplant:
  Plerixafor (AMD3100) Starting dose of 0 (escalating doses 80, 160, 240 mcg/kg) given daily subcutaneously in abdomen for 4 doses + Thymoglobulin (ATG) 0.5 mg/kg on day -3; 1.5 mg/kg on day -2; & 2 mg/kg on day -1. Given only to patients with unrelated donors + G-CSF (Filgrastim) 10 mcg/kg subcutaneous injection beginning on day -9 daily for 6 days + Fludarabine 40 mg/m^2 beginning on Day -6 for four consecutive days + Busulfan 130 mg/m^2 for four consecutive days, immediately after completion of Fludarabine + Allogeneic blood stem cell transplant of Stem Cell Infusion (Bone marrow or PBPC)
Arm/Group | Phase I Plerixafor + G-CSF | Phase II Plerixafor 240 mcg/kg + G-CSF
Serious Adverse Events (participants affected / at risk) | 8/18 | 6/29
Other Adverse Events (participants affected / at risk) | 17/18 | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Plerixafor + G-CSF (N=18) | Phase II Plerixafor 240 mcg/kg + G-CSF (N=29)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neutropenic fever (Infections and infestations) | 1 (1) | 0 (0)
Hemorrhagic cyctitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Central Nervous System (CNS) hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 3 (4) | 4 (4)
Fall (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Death (General disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — with Cytomegalovirus (CMV)
Graft versus Host Disease, Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Plerixafor + G-CSF (N=18) | Phase II Plerixafor 240 mcg/kg + G-CSF (N=29)
Elevated White Blood Count (Blood and lymphatic system disorders) | 8 (8) | 11 (12)
High Blood Pressure (Cardiac disorders) | 5 (6) | 4 (4)
Change in cardiac function (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 9 (25) | 5 (5)
Nausea (Gastrointestinal disorders) | 7 (9) | 15 (16)
Dysphagia (Gastrointestinal disorders) | 8 (9) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 6 (6)
Flu-like Symptoms (General disorders) | 12 (17) | 15 (15) — Fever, chills
Alkaline phosphatase Increase (Investigations) | 14 (14) | 4 (4)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Infections (Infections and infestations) | 16 (36) | 11 (17)
Metabolism and nutrition disorders: Changes within blood level (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2)
Nervous system disorders (Nervous system disorders) | 8 (10) | 3 (3)
Urinary changes (Renal and urinary disorders) | 1 (1) | 0 (0)
Hemoglobinuria (Renal and urinary disorders) | 1 (1) | 3 (3)
Genitourinary disorders (Renal and urinary disorders) | 5 (6) | 2 (2)
Respiratory Infection, Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 9 (16) | 10 (13)
Graft versus Host Disease (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No